CLINICAL TRIAL: NCT05520008
Title: A Game-based Foot & Ankle Exercise Program to Increase Efficacy Of Compression Garments At Managing Edema
Brief Title: Game-Based Foot & Ankle Exercise for Those With Lower Extremity Edema
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: Medline Industries (Industry)
Responsible Party: Principal Investigator, Bijan Najafi, PhD, Professor of Surgery, Baylor College of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: H-52182
Record Dates: First submitted 2022-08-26; First posted 2022-08-29 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Lower Extremity Swelling; Lower Extremity Edema; Venous Insufficiency of Leg
Keywords: Compression Garment; Game-based Exercise

STUDY DESIGN:
Intervention Model Description: Participants who satisfy the inclusion and exclusion criteria and sign the informed consent form will be randomly assigned with a ratio of 1:1 into two groups. Both groups will be given a compression garment (CompreCares, Medline, IL, USA) to wear for the 4 weeks of the study. The Active group (AG) will also be allocated a tablet and foot sensor so that they can play game-based foot & ankle exercises during the same time period. The other group (Control group, CG) will only use the compression garment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active group (AG) (Experimental): Active group (AG). The AG (n=15) will play game-based foot and ankle exercises via a mobile application on a tablet. They will be asked to wear a foot sensor that is connected to the tablet during the exercise. They will be asked to play the game for 5-minutes, daily. They will do this in conjunction with wearing a compression garment for a period of 4 weeks.
  Interventions: Other: Game-based exercise
- Control group (CG) (No Intervention): Control Group (CG). The CG (n=15) will wear a compression garment for four weeks.

INTERVENTIONS:
Other: Game-based exercise — Patients in the active group will put on a sensor connected to a tablet to play a game-based foot/ankle exercise twice a day for 5 minutes for four weeks.
  Other Names: Tele-exercise
  Arms: Active group (AG)

SUMMARY:
The present study aims to use a game-based tele-exercise program for patients using a compression garment to improve lower extremity edema. This tele-exercise gaming platform can work as an efficient exercise to improve patients' muscle strength. It also can be helpful in improving edema and venous return and can be used in addition to compression garments to increase efficacy. The sample size (n=30) is convenient and designed to explore acceptability and feasibility. Eligible participants will be screened at the Baylor college of Medicine Clinic based on the inclusion/exclusion criteria. Participants who satisfy the inclusion and exclusion criteria and sign the informed consent form will be randomly assigned with ratio of 1:1 into two groups. Both groups will receive a compression garment to use for 4 weeks, and in the intervention group, patients will receive a sensor and a tablet to play foot & ankle exercise games twice a day for 5 minutes. Study participation will be 4 weeks for all participants. Participants will be assessed in two visits: a baseline visit (BL) and a visit at the end of the 4 weeks (W4). The primary outcomes will be calf circumference, foot volume, and pitting edema grade. Secondary outcomes include limb strength, foot perfusion, gait assessment (gait speed, stride length, double stance, and gait steadiness), balance, and quality of life. The coordinator will monitor patients weekly to see their adherence to the compression garment and game-based exercise.

DETAILED DESCRIPTION:
Lower extremity edema (LE) is an accumulation of interstitial fluid volume in the legs and feet and commonly occurs in patients with diabetes, hypertension, kidney disease, heart failure, cirrhosis, cancer, and obesity. LE can also result from deep vein thrombosis (DVT) in the lower leg. Compression socks or garments are often used to decrease this edema. Despite the efficacy of this treatment, there are some limitations including low patient compliance and contraindication of high compression levels for patients with high grades of peripheral arterial disease. Given that it is has previously been shown that exercise can be a positive way to reduce LE, the present study aims to use a game-based exercise program to help increase patient's movement and thus improve efficacy and adherence to the compression garments/socks.

The investigators will recruit 30 participants and randomly divide them into two groups: Active Group (AG) and Control Group (CG). Both groups will receive a compression garment (CompreCares) developed by Medline Incorporated(Inc). (IL, USA). The AG will receive a tablet and foot sensor (TEXASSENSE INC, USA), and will be instructed to play with it daily for 5 minutes over the period of 4 weeks.

During the two study visits (BL and W4), the investigators will assess the following outcomes: calf muscle activation (assessed by surface electromyography [sEMG]), foot perfusion (SNAPSHOT NIR, Kent Imaging System), calf and foot circumference, ankle-brachial index (ABI), pitting edema test, foot volume, gait, balance, and peripheral neuropathy (DPNCheck, Neurometrix Inc., Woburn, Massachusetts, USA).

Acceptability and patient reported outcomes will be assessed via validated questionnaires collected at each study visit.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (18+ years old) who have lower extremity edema
* Willing to attend clinic for assessments

Exclusion Criteria:

* Severe cognitive decline that reduces their ability to use tele-foot exercise device
* Major visual problems that reduces their ability to use tele-foot exercise device
* Inability to walk independently for a distance of 10 meters
* Major foot problems such as active lower extremity wounds
* Major foot deformity (e.g., Charcot Foot)
* Previous major amputations, and claudication
* Decompensated or advanced heart failure New York Heart Association (NYHA) Functional Class(FC) III-IV
* Significant heart disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2022-11-03 (Actual); Primary Completion 2023-10-06 (Actual); Study Completion 2023-10-06 (Actual)

PRIMARY OUTCOMES:
Change in calf circumference from baseline to 4 weeks | 4 weeks from baseline
  Calf circumference will be assessed with a soft measuring tape for each leg
Change in foot circumference from baseline to 4 weeks | 4 weeks from baseline
  Foot circumference will be assessed with a soft measuring tape for each leg
Change in foot volume from baseline to 4 weeks | 4 weeks from baseline
  Foot volume will be assessed with a standard foot volumeter
Change in pitting edema grade from baseline to 4 weeks | 4 weeks from baseline
  Coordinators will press on the affected area in the lower extremities and measure depth of indention. They will record the length of skin rebound time and grade the edema based on validated scales

SECONDARY OUTCOMES:
Change in gastrocnemius muscle strength from baseline to 4 weeks | 4 weeks from baseline
  Lower extremity strength will be assessed with an ankle dynamometer and surface electromyography (Delsys Trigno Wireless EMG System, MA, US).
Change in gait and balance from baseline to 4 weeks | 4 weeks from baseline
  Gait speed will be measured with standard walking tests and wearable sensors (Legsys).
Change in balance from baseline to 4 weeks | 4 weeks from baseline
  Static balance will be measured with standard balance tests and wearable sensors (Balansens).
Change in plantar tissue oxygen saturation/consumption from baseline to 4 weeks | 4 weeks from baseline
  Percentage of tissue oxygen saturation (SatO2) and hemoglobin values will be measured using a validated near-infrared (NIR) camera (Snapshot NIR, KENT Imaging Inc., Calgary, AB, Can) that detects an approximate value of real-time SatO2 and level in superficial tissue. The area that will be captured is the metatarsus area

OTHER OUTCOMES:
Change in peripheral neuropathy from baseline to 4 weeks | 4 weeks from baseline
  Peripheral neuropathy will be assessed using DPNCheck (Neurometrix, Woburn, MA, USA). This is a noninvasive device which will measure conduction velocity and amplitude.
Patient acceptance at 4 weeks | 4 weeks from baseline
  Participant acceptance of the tele-exergaming program will be assessed at the end of their participation using a validated technology acceptance model (TAM) questionnaire
Change in physical activity (step count and intensity minutes) from baseline to 4 weeks | 4 weeks from baseline
  Physical activity metrics, such as step count and intensity minutes, will be measured over the course of the 4 weeks using a smart watch (Vivosmart 4, Garmin, US)

CONTACTS AND LOCATIONS:
Overall Officials: Bijan Najafi, PhD, Principal Investigator — Baylor College of Medicine
Locations (1):
- Baylor College of Medicine, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No